CLINICAL TRIAL: NCT04613479
Title: Frequency of Hepatobilliary Manifestations in Patients With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hayam Fathy Nasr, clinical doctor internal medicine, Assiut University
Other Study IDs: Inflammatory bowel disease
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Hepatobilliary Manifestations in Inflammatory Bowel Disease Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatobilliary manifestations as extraintestinal manifestations of IBD are sometimes underdiagnosed which can impair patient prognosis

DETAILED DESCRIPTION:
Non alcoholic fatty liver is aliver disease most commonly found in patient with IBD most commonly without intestinal activity.

On the other hand primary according cholangitis is the most common specific with IBD commonly with ulcerative colitis. and is commonly overlap with autoimmune hepatitis IBD therapy can also be a cause it can lead to hepatic toxicity and some drugs like ant TNF can cause hepatitis b virus activation.

ELIGIBILITY:
Inclusion Criteria:all patients diagnosed IBD crohns and ulcerative on conventional treatment and biological treatment -

Exclusion Criteria:no

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients diagnosed IBD either crohns or ulcerative, male or female, age above 18 years old.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The prevelance of hepatobilliary manifestations in IBD patients | 1 year